CLINICAL TRIAL: NCT00499473
Title: A Pharmacokinetic and Phase 2 Study of Sunitinib Malate in Recurrent Malignant Gliomas
Brief Title: Sunitinib in Treating Patients With Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00215; NCI-2009-00215 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-IRB-2006C0098; CDR0000554443; OSU-06060; OSU 06060 (Other: Ohio State University Medical Center); 7745 (Other: CTEP); N01CM62207 (NIH); N01CM62203 (NIH); P30CA016058 (NIH); N01CM62206 (NIH)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Diffuse Astrocytoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Adult Oligodendroglioma; Adult Pineal Gland Astrocytoma
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Gliosarcoma; Glioma; Oligodendroglioma | interventions — Sunitinib

ARMS (2):
- Stratum 1 (kinase inhibitor therapy) (Experimental): Non-EIAC patients receive oral sunitinib malate once daily for 4 consecutive weeks followed by 2 weeks of rest.
  Interventions: Drug: sunitinib malate; Other: pharmacological study
- Stratum 2 (kinase inhibitor therapy) (Experimental): EIAC & OSU patients receive oral sunitinib malate as in stratum 1. Patients receive escalating doses of oral sunitinib malate until the maximum tolerated dose (MTD) is determined.
  Interventions: Drug: sunitinib malate; Other: pharmacological study

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU11248; sunitinib; Sutent
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial is studying how well sunitinib works in treating patients with recurrent malignant gliomas. Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of sunitinib malate in patients with recurrent malignant gliomas as measured by 6-month progression-free survival.

II. To determine the lower of the dose of sunitinib malate in patients receiving enzyme-inducing anti-convulsants that would achieve similar serum drug and metabolite concentrations as that in patients not receiving enzyme-inducing anticonvulsants or the maximum tolerated dose in the same population.

SECONDARY OBJECTIVES:

I. To examine the toxicity and safety of sunitinib malate in patients with the above noted tumors.

II. To evaluate tumor responses in the stated patients. III. To evaluate progression-free and overall survival in the stated patients.

OUTLINE: This is a multicenter study. Patients are stratified according to use of enzyme-inducing anticonvulsants (EIAC) (yes vs no).

STRATUM 1 (non-EIAC): Patients receive oral sunitinib malate once daily for 4 consecutive weeks followed by 2 weeks of rest.

STRATUM 2 (EIAC & OSU patients only): Patients receive oral sunitinib malate as in stratum 1. Patients receive escalating doses of oral sunitinib malate until the maximum tolerated dose (MTD) is determined.

Patients undergo blood sample collection periodically for pharmacokinetic studies. Samples are analyzed for plasma concentrations of sunitinib malate via LC/MS/MS method.

In both strata, treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Stratum 1:

  * Currently not receiving an enzyme-inducing anticonvulsant

    * Patients receiving non-enzyme inducing anticonvulsants are eligible for this stratum
  * Histologically confirmed WHO grade IV astrocytoma (glioblastoma multiforme [GBM]) including gliosarcoma
* Stratum 2 (USA patients only):

  * Currently on stable dose of an enzyme-inducing anticonvulsant (with confirmed therapeutic serum levels) for at least 2 weeks prior to study registration including any of the following:

    * Phenytoin
    * Carbamazepine
    * Phenobarbital
  * Histologically confirmed grade IV astrocytoma (GBM), gliosarcoma, grade III astrocytoma, oligodendroglioma, or mixed oligoastrocytoma
* All patients must have unequivocal evidence of tumor progression by MRI or CT scan performed no longer than 14 days prior to study registration

  * Patients undergoing surgery for progressive disease with nonmeasurable disease on post-operative MRI, ideally obtained within 48 hours of surgery, (i.e., macroscopic gross total resection) are eligible
* ECOG performance status 0-2 (Karnofsky ≥ 60%)
* Life expectancy > 3 months
* Leukocytes ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9 g/dL
* Serum calcium ≤ 12.0 mg/dL
* Total bilirubin within normal institutional limits (ULN)
* AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional ULN
* Creatinine < 1.5 X institutional ULN
* Patients must have QTc < 500 msec
* The following groups of patients are eligible provided they have New York Heart Association class II cardiac function on baseline ECHO or MUGA:

  * Those with a history of class II heart failure who are asymptomatic on treatment
  * Those with prior anthracycline exposure
  * Those who have received central thoracic radiation that included the heart in the radiotherapy port
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation

  * All women of childbearing potential must have a negative pregnancy test prior to receiving sunitinib malate
* Patients with a history of QTc prolongation (defined as a QTc interval >= 500 msec), serious ventricular arrhythmia (VT or VF > 3 beats in a row) or other significant ECG abnormalities are excluded
* Patients with poorly controlled hypertension (systolic BP ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg) are ineligible
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain sunitinib malate tablets are excluded
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
  * History of myocardial infarction, cardiac arrhythmia, stable or unstable angina, symptomatic congestive heart failure, or coronary or peripheral artery bypass graft or stenting within 12 months prior to study entry
  * Class III or IV heart failure as defined by the NYHA functional classification system
* Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medication are ineligible
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infections requiring antibiotics or psychiatric illness/social situations that would limit compliance with study requirements are ineligible
* Pregnant women are excluded from this study
* Breastfeeding should be discontinued if the mother is treated with sunitinib malate
* Patients are eligible if they received up to 1 previous chemotherapy regimen
* ≥ 12 weeks must have elapsed from the completion of radiation therapy
* ≥ 4 weeks from previous non-nitrosoureas-based cytotoxic chemotherapy
* ≥ 6 weeks from any nitrosoureas
* ≥ 2 weeks from last cytostatic chemotherapy such as erlotinib hydrochloride or tamoxifen
* Patients who have undergone previous stereotactic radiosurgery, intratumoral chemotherapy, or brachytherapy are eligible if functional imaging (PET or SPECT scan, MR spectroscopy, or dynamic MRI) supports the diagnosis of recurrent tumor or recurrent disease is confirmed histologically
* Concurrent steroids allowed provided the patients is on a stable or decreasing dose for at least 7 days prior to baseline tumor assessment (MRI and/or CT scan)
* Patients who have received prior treatment with any other antiangiogenic agent (e.g., bevacizumab, sorafenib, pazopanib, AZD2171, PTK787, or VEGF Trap) are ineligible
* Patients who require use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin or enoxaparin are excluded, although warfarin doses of up to 2 mg daily are permitted for prophylaxis of thrombosis

  * Low molecular weight heparin is permitted provided the patient's PT INR is < 1.5
* Use of agents with proarrhythmic potential (e.g., terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, or flecainide) is not permitted during the study
* No other investigational or commercial agents or non-investigational therapy designed to treat the brain malignancy (i.e., radiation therapy, systemic or intratumoral chemotherapy, biological agents, immunotherapy, or hormonal therapy) is allowed during the study period
* HIV-positive patients on combination antiretroviral therapy are ineligible

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biological composition to sunitinib malate
* Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or radiation therapy within 12 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier

  * At least 4 weeks must have elapsed since any major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cavaliere, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum I: Non-EIAC: Patients will take one 50-mg capsule of sunitinib orally once daily for 4 consecutive weeks followed by 2 weeks of rest (drug holiday) with no sunitinib.
- Stratum 2: EIAC: The first six patients enrolled on stratum 2 will be dosed identical to those patients on stratum 1.The dosage of the next 6-patient cohort in stratum 2 will be adjusted to that predicted by pharmacokinetic modeling to provide the same concentrations seen in first six non-enzyme inducing patients.
Period: Overall Study
Arm/Group | Stratum I: Non-EIAC | Stratum 2: EIAC
Started | 27 | 4
Completed | 21 (Patients evaluable) | 4
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stratum I: Patients Not on EIAC: Patients will take one 50-mg capsule of sunitinib orally once daily for 4 consecutive weeks followed by 2 weeks of rest (drug holiday) with no sunitinib.
- Stratum 2: Patients on EIAC: The first six patients enrolled on stratum 2 will be dosed identical to those patients on stratum 1.The dosage of the next 6-patient cohort in stratum 2 will be adjusted to that predicted by pharmacokinetic modeling to provide the same concentrations seen in first six non-enzyme inducing patients.
- Total: Total of all reporting groups
Arm/Group | Stratum I: Patients Not on EIAC | Stratum 2: Patients on EIAC | Total
Number analyzed (Participants) | 27 | 4 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 4 | 25
  >=65 years | 6 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 0 | 11
  Male | 16 | 4 | 20
Region of Enrollment [Number; unit: participants]
  United States | 27 | 4 | 31

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months (Stratum 1)
Description: Number of patients with Progression-free Survival at 6 months for Stratum 1
Time Frame: From time to registration to up to 6 months
Population: Only 21 patients were evaluable for PFS
Measure: Number; unit: patients
Arm/Group | Stratum I: Non-EIAC | Stratum 2: EIAC
Number analyzed (Participants) | 21 | 0
patients | 1 |

2. Primary Outcome: Maximum Tolerable Dose Based on Dose-limiting Toxicity of Sunitinib in Patients Receiving EIAC (Stratum 2)
Description: Maximum tolerable dose of sunitinib in patients receiving treatment with EIAC agents using dose escalation based on the steady-state trough sunitinib + SU12662 plasma concentrations on day 14 observed in patients treated in stratum 1. Six patients will be treated in each dose cohort with up to 12 patients being treated at the maximum tolerable dose for a total of 18-24 patients with gliomas receiving EIAC.
Time Frame: From the time of first treatment with sunitinib until completion of treatment, assessed up to 30 days
Population: MTD in Stratum 2 not determined due to lack of efficacy in Stratum 1
Arm/Group | Stratum I: Non-EIAC | Stratum 2: EIAC
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Dose Resulting in Steady-state Trough
Description: Average of pre-dose values of sunitinib + SU12662 plasma concentrations equivalent to that observed in patients not receiving EIAC based on pharmacokinetic modeling.
Time Frame: At baseline (day 8) and days 15, 22, and 23
Population: Not determined due to early termination of the study due to lack of efficacy
Arm/Group | Stratum I: Non-EIAC | Stratum 2: EIAC
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Confirmed Objective Response (Complete Response[CR] or Partial Response [PR])
Description: Confirmatory scans should also be obtained within 4 to 6 weeks following initial documentation of objective response. Confidence intervals for the true proportion will be calculated using the exact binomial method. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to 12 weeks
Population: Only 21 patients were evaluable for response
Measure: Number; unit: patients
Arm/Group | Stratum I: Non-EIAC | Stratum 2: EIAC
Number analyzed (Participants) | 21 | 4
patients
  Complete Response Rate | 0 | 0
  Partial Response Rate | 0 | 0

5. Secondary Outcome: Percentage of Patients Progression Free at 12 Months
Time Frame: At 12 months after the start of treatment
Measure: Number; unit: percent of patients
Arm/Group | Stratum I: Non-EIAC | Stratum 2: EIAC
Number analyzed (Participants) | 21 | 4
percent of patients | 0 | 0

6. Secondary Outcome: Overall Survival
Time Frame: up to 12 months
Measure: Median (Full Range); unit: months
Arm/Group | Stratum I: Non-EIAC | Stratum 2: EIAC
Number analyzed (Participants) | 27 | 4
months | 5.7 [2.9 to 29.9] | 12.3 [3.3 to 15.6]

ADVERSE EVENTS:
Description: The NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 was utilized for Adverse event reporting.
Groups:
- Stratum 2: EIAC: Patients will take one 50-mg capsule of sunitinib orally once daily for 4 consecutive weeks followed by 2 weeks of rest (drug holiday) with no sunitinib. In addition to EIAC (Enzyme-inducing anticonvulsant)
Arm/Group | Stratum I: Non-EIAC | Stratum 2: EIAC
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/4
Other Adverse Events (participants affected / at risk) | 27/27 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum I: Non-EIAC (N=27) | Stratum 2: EIAC (N=4)
Alanine aminotransferase increased (Investigations) | 5 (6) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Blurred vision (Eye disorders) | 2 (2) | 1 (1)
Confusion (Psychiatric disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 9 (10) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 7 (11) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Fatigue (Gastrointestinal disorders) | 11 (14) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 2 (6) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Hypertension (Vascular disorders) | 4 (5) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) — right and left sided
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nervous system disorder (Nervous system disorders) | 3 (3) | 0 (0) — Imbalance, nystagmus
Neutrophil count decreased (Investigations) | 5 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Neuropathy (Nervous system disorders) | 4 (4) | 1 (1) — sensory and motor
Platelet count decreased (Blood and lymphatic system disorders) | 3 (5) | 2 (2)
Pyramidal tract syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 2 (2)
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Vascular disorder (Vascular disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
White blood cell decreased (Investigations) | 5 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less